CLINICAL TRIAL: NCT06217627
Title: The Potential of Umbilical Cord Stem Cell Secretions in Skin Rejuvenation
Brief Title: Skin Rejuvenation Using Stem Cell Secretome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: COR clinic of Regenerative Medicine (Network)
Responsible Party: Principal Investigator, Nada Alaaeddine, Dean of health Sciences at MUBS, Modern University for Business and Science
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2021-cor001
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Skin Rejuvenation
MeSH Terms: interventions — Secretome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical cord (UC)- mesenchymal stem cells (MSCs) secretome (Experimental): 19 participants received UC-MSCs secretome injections in the neck and different areas of the face including the forehead, cheeks, under eyes, chin, and nasolabial folds.
  Interventions: Biological: secretome
- UC-explants secretome (Experimental): 30 participants received UC-explants secretome in the left and right hands
  Interventions: Biological: secretome

INTERVENTIONS:
Biological: secretome — The secretome is the secretions of MSCs or explants from umbilical cord tissues. It contains diverse trophic molecules including cytokines, chemokines, angiogenic factors, and growth factors.

SUMMARY:
This clinical trial aims to investigate the effect of umbilical cord explants (UC)-explants and UC-mesenchymal stem cells (MSCs) secretome on skin rejuvenation, to provide future reference or standard in the application of cell free-based therapy in skin aging.

DETAILED DESCRIPTION:
This trial is a pilot clinical trial evaluating the effect of the secretions of umbilical cord explants and mesenchymal stem cells on skin rejuvenation. Also the concentration of selected growth factors was assessed in the secretome derived from UC-explants and UC-MSCs.

Healthy women participants, after their consent, received secretome injections in their hands, face, and neck. Outcomes were assessed on the Hand Volume Rating Scale, Wrinkle Severity Rating Scale, and through histologic examination of skin biopsy at two different times: before treatment and after 12 months. A digital camera was used to obtain photographs of hands, face, and Neck at each visit. These were assessed by a single-blinded dermatologist. SPSS software version 26 (64-bit) was used for all analyses.

Participants provided written informed consent and were asked not to change their routine skin care habits during the study.

ELIGIBILITY:
Inclusion Criteria:

* women participants aged > 25 years
* any skin type according to the Glogau scale
* Willing to be a research subject, sign a consent form, and commit to follow-up visits

Exclusion Criteria:

* patients with active skin diseases (e.g. atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis)
* patients using other anti-aging treatments within 1 month

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the fact that women are more likely than men to keep track of their skin condition more regularly and to adhere to study procedures, women participants were chosen in this study to homogenize the data and prevent drop-outs.
Enrollment: 49 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Selected growth factors assessment | 4 samples of secretome extracted from UC-explants with one week interval. 1 sample of secretome extracted from confluent UC-MSCs at passage 1
  assessment of the concentration (pg/ml) of selected growth factors (bFGF, HGF, TIMP-3, VEGF, andTGF-b) in the secretome derived from UC-explants and UC-MSCs using ELISA essays.
Wrinkle severity in hands | digital photographs before injection and after 7 months.
  wrinkle severity was assessed in the hands by the Hand Volume Rating Scale: grade 0 (absent) to grade 4 (severe)
Wrinkle severity in the face and neck | digital photographs before injection and after 7 months.
  wrinkle severity was assessed by the Wrinkle Severity Rating Scale: grade 0 (no wrinkles) to grade 5 ((very deep wrinkle and redundant fold)

SECONDARY OUTCOMES:
Histological examination | skin biopsies were performed at two moments: before treatment and after 12 months.
  The histological examination of skin biopsies evaluated the assessment of collagen, keratin, elastin, basement membrane of blood vessels, and fibroblast nuclei.

CONTACTS AND LOCATIONS:
Overall Officials: Nada Alaaeddine, PhD, Principal Investigator — COR clinic of Regenerative Medicine
Locations (1):
- COR clinic of Regenerative Medicine, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No